CLINICAL TRIAL: NCT02253147
Title: A Controlled, Randomized, Double-Blinded, Within-Subject, Multicenter, Prospective Clinical Study of TEOSYAL® RHA (Resilient Hyaluronic Acid) Ultra Deep Versus Perlane-L® in the Treatment of Moderate to Severe Nasolabial Folds
Brief Title: TEOSYAL® RHA Ultra Deep and Perlane-L® for the Correction of Nasolabial Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teoxane SA (Industry)
Collaborators: ethica Clinical Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TEO-RHA-1402
Record Dates: First submitted 2014-09-25; First posted 2014-10-01 (Estimated); Results first posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-02

CONDITIONS: Nasolabial Folds, Wrinkles
Keywords: Nasolabial folds; Dermal filler; Hyaluronic acid (HA); Wrinkles

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Left side TEOSYAL® RHA Ultra Deep, Right side Perlane-L® (Experimental): Split-face injection of TEOSYAL® RHA Ultra Deep into the left Naso Labial Folds (NLFs) and Perlane-L® into the right NLF (n=120). Up to 3.0 mL injected per NLF. Touch-up treatment provided at 2 weeks (up to 3.0 mL per NLF).
  Interventions: Device: TEOSYAL® RHA Ultra Deep
- Left side Perlane-L®, Right side TEOSYAL® RHA Ultra Deep (Experimental): Split-face injection of Perlane-L® into the left Naso Labial Folds (NLFs) and TEOSYAL® RHA Ultra Deep into the right NLF (n=120). Up to 3.0 mL injected per NLF. Touch-up treatment provided at 2 weeks (up to 3.0 mL per NLF).
  Interventions: Device: TEOSYAL® RHA Ultra Deep

INTERVENTIONS:
Device: TEOSYAL® RHA Ultra Deep — A sterile, biodegradable, biocompatible, viscoelastic, clear, colorless, homogenized gel implant. It consists of cross-linked hyaluronic acid produced by fermentation of Streptococcus equi bacteria, formulated to a concentration of 23 mg/mL and 0.3% w/w lidocaine in a physiologic buffer. It is supplied in individual treatment syringes with 27Gauge ½" disposable sterile needles.

SUMMARY:
The purpose of this study is to compare the effectiveness and safety of TEOSYAL® RHA Ultra Deep versus Perlane-L® in the treatment of moderate to severe nasolabial folds. This is a controlled, randomized, double-blinded, within subject (split-face), multicenter, prospective clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, male or female of any race, 22 years of age or older; female subjects of childbearing potential must have a negative Urine Pregnancy Test and practice a reliable method of contraception;
* NLFs classified as WSRS grade 3 or 4 (same score for each side);
* Willing to abstain from facial aesthetic procedures/therapies that could interfere with study evaluations;
* Able to follow study instructions and likely to complete all required visits;
* Signed informed consent and HIPAA form.

Exclusion Criteria:

* Female subjects that are pregnant, breast-feeding or of childbearing potential and not practicing reliable birth control;
* Known hypersensitivity/allergy to any component of the study devices;
* Known sensitivity to local anesthetics of the amide type, history of multiple severe allergies, history of anaphylactic shock;
* Known susceptibility to keloid formation, hypertrophic scarring or clinically significant skin pigmentation disorders;
* Clinically significant active skin disease within 6 months;
* History of active chronic debilitating systemic disease;
* History of connective tissue disease;
* History of malignancy (excl. non-melanoma skin cancer) within past 5 years;
* History of bleeding disorders;
* Need for clinically significant and continuous medical treatment within 2 weeks prior to first visit;
* Received/used a prohibited treatment/procedure within certain time periods (e.g., bioresorbable fillers, NSAIDS, ASA, high dose vitamin E, corticosteroids, interferon, anti-coagulation therapies, laser/light therapies, botulinum toxin injections (frontalis and glabella complex treatment permitted), prescription strength topical retinoids, facial peels, excisional facial surgery, clinically significant oral or maxillofacial surgery).
* Evidence of clinically significant alcohol or drug abuse, or history of poor cooperation, non-compliance with medical treatment, or unreliability
* Exhibit a physical attribute(s) that may prevent assessment or treatment of NLFs such as excessive facial hair, traumatic or surgical facial scars, and/or excessive hyperpigmentation in the treatment areas.
* A condition or situation that may put the subject at significant risk, confound the study results, or significantly interfere with the subject participation.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - United States, Beverly Hills, California
  - United States, Bradenton, Florida
  - United States, Chapel Hill, North Carolina
  - United States, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 120 were randomized for a split-face injection of RHA Ultra Deep and Perlane-L.
  20 subjects were randomized to an untreated group (recruited only to avoid Blinded Live Evaluator to be biased so, not presented)
Pre-assignment Details: 2 subjects randomized to the RHA UD/Perlane discontinued participation prior to receiving study treatment (N=118) 2 subjects randomized to the untreated group received injections with RHA UD/Perlane. These subjects were placed in the SAFT population for safety evaluations (SAFT population n=120)
Groups:
- TEOSYAL® RHA Ultra Deep / Perlane-L®: Split-face injection of TEOSYAL® RHA Ultra Deep into one NLF and Perlane-L® into the contralateral NLF. Up to 3.0 mL injected per NLF (deep-dermis to superficial subcutaneous). Touch-up treatment provided at 2 weeks (up to 3.0 mL per NLF).
  TEOSYAL® RHA Ultra Deep: A sterile, biodegradable, biocompatible, viscoelastic, clear, colorless, homogenized gel implant. It consists of cross-linked hyaluronic acid produced by fermentation of Streptococcus equi bacteria, formulated to a concentration of 23 mg/mL and 0.3% w/w lidocaine in a physiologic buffer. It is supplied in individual treatment syringes with 27G½" disposable sterile needles.
Period: Overall Study
Arm/Group | TEOSYAL® RHA Ultra Deep / Perlane-L®
Started | 118
N Patients at W24 (Primary Outcome) | 88
N Patients at W36 | 86
N Patients at W52 | 84
Completed (N patients completed W64) | 71
Not Completed | 47
Not completed — Protocol Violation | 30
Not completed — Did not consent to study extension | 9
Not completed — Conditional re-treatment at W52 | 5
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | TEOSYAL® RHA Ultra Deep / Perlane-L®
Number analyzed (Participants) | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30
  Not Hispanic or Latino | 88
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 97
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 118
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — The Fitzpatrick scale is a numerical classification schema for human skin color.
  Type I - always burns, never tans (pale white; blond or red hair; blue eyes; freckles).
  Type II - usually burns, tans minimally (white; fair; blond or red hair; blue, green, or hazel eyes) Type III - sometimes mild burn, tans uniformly (cream white; fair with any hair or eye color) Type IV - burns minimally, always tans well (moderate brown) Type V - very rarely burns, tans very easily (dark brown) Type VI - Never burns, never tans (deeply pigmented dark brown to darkest brown)
  Participants
    Types I to III | 65
    Types IV to VI | 53

OUTCOME MEASURES:

1. Primary Outcome: Non-inferiority of the Delta of the WSRS Score Between W24 and Baseline for TEOSYAL® RHA Ultra Deep Versus Perlane-L® for the Correction of Moderate to Severe Naso-Labial Folds Based on the Wrinkle Severity Rating Scale (WSRS) Score Assessed by the BLE.
Description: WSRS (Wrinkle Severity Rating Scale) is a validated 5-point scale with 1 being 'absent' and 5 being 'extreme'.
  BLE =Blinded Live Evaluator
Time Frame: Baseline and 24 weeks after last treatment
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- TEOSYAL® RHA Ultra Deep: Injection of TEOSYAL® RHA Ultra Deep into one NLF
- Perlane-L®: Injection of Perlane-L® into the controlateral NLF
Arm/Group | TEOSYAL® RHA Ultra Deep | Perlane-L®
Number analyzed (Participants) | 88 | 88
units on a scale | -1.34 [-1.46 to -1.22] | -1.16 [-1.29 to -1.03]
Statistical Analysis 1: Comparison: TEOSYAL® RHA Ultra Deep vs Perlane-L®; Efficacy of TEOSYAL® RHA Ultra Deep versus control is analyzed in a non-inferiority statistical model using the 5-grade Wrinkle Severity Rating Scale (WSRS) as rated by the Blinded Live Evaluator at 24 weeks after baseline. The primary endpoint is the aesthetic improvement from pre-injection of the NLF at the side of the face treated with TEOSYAL® RHA Ultra Deep compared to the one at the side of the face treated with the control device, as assessed by the BLE at 24 weeks after baseline; Test type: Non-Inferiority — A WSRS change of 1 grade is considered to be clinically significant. A difference of ≤0.5 grade between the two treatment groups (i.e., half of the clinically significant difference) = non-inferiority margin. The primary efficacy endpoint uses a paired-design and is analyzed by calculating two-sided confidence intervals of the mean difference between TEOSYAL® RHA UD and the control device, between the V1 enrollment visit (baseline) and V7 (24 weeks after baseline); Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.34 to -0.11] — The decision is based on the upper limit of the 2-sided confidence interval for the difference for the change from baseline, between test and comparator treatment. For achieving non-inferiority, the upper confidence limit of a 95.0% CI must be ≤0.5

2. Secondary Outcome: Post Injection Treatment Responses (From Common Treatment Responses (CTR) Diary) for Safety Evaluation of TEOSYAL® RHA Ultra Deep Versus Perlane-L®
Description: The subjects received a diary booklet and instructions for recording his/her observations of the Common Treatment Responses of the study treatments for the first 14 days after each treatment (initial, touch-up). The diary was discussed during each telephone follow-up visit. Subjects should complete the diary at approximately the same time each day (i.e., am or pm).
  The subject diary captured the following Common Treatment Responses (CTR) that occur following the injection of a dermal filler; specifically, redness, pain, tenderness, firmness, swelling, lumps/bumps, bruising, itching, discoloration, and "other".
  The 14-day patient CTR diary included a detailed glossary describing all signs/symptoms listed in the diary; an option was provided to rate "other" if the subject experienced a sign/symptom that is not listed.
  The table presents the number of subjects experiencing at least 1 Common Treatment Response (CTR)
Time Frame: During 14 days after initial treatment (D0) and touch-up (2 weeks)
Population: CTR are presented for the SAFT population (N=120) (see pre-assignment details) Number of patients for CTR after touch-up treatment are based on number of patients receiving Touch-up treatment (RHA-UD N=32/Perl N=47)
Measure: Count of Participants; unit: Participants
Arm/Group | TEOSYAL® RHA Ultra Deep | Perlane-L®
Number analyzed (Participants) | 120 | 120
Participants
  Bruising (initial treatment) | 70 | 72
  Bruising (Touch-up): number analyzed (Participants) | 32 | 47
  Bruising (Touch-up) | 17 | 22
  Discolouration (initial treatment) | 50 | 56
  Discolouration (Touch-up): number analyzed (Participants) | 32 | 47
  Discolouration (Touch-up) | 9 | 12
  Firmness (initial treatment) | 91 | 93
  Firmness (Touch-up): number analyzed (Participants) | 32 | 47
  Firmness (Touch-up) | 24 | 36
  Itching (initial treatment) | 30 | 44
  Itching (Touch-up): number analyzed (Participants) | 32 | 47
  Itching (Touch-up) | 4 | 10
  Lumps/Bumps (initial treatment) | 81 | 90
  Lumps/Bumps (Touch-up): number analyzed (Participants) | 32 | 47
  Lumps/Bumps (Touch-up) | 18 | 30
  Pain (initial treatment) | 66 | 87
  Pain (Touch-up): number analyzed (Participants) | 32 | 47
  Pain (Touch-up) | 16 | 31
  Redness (initial treatment) | 84 | 91
  Redness (Touch-up): number analyzed (Participants) | 32 | 47
  Redness (Touch-up) | 17 | 31
  Swelling (initial treatment) | 97 | 104
  Swelling (Touch-up): number analyzed (Participants) | 32 | 47
  Swelling (Touch-up) | 27 | 38
  Tenderness (initial treatment) | 90 | 95
  Tenderness (Touch-up): number analyzed (Participants) | 32 | 47
  Tenderness (Touch-up) | 21 | 35

3. Secondary Outcome: Assessment of Injection Site Pain (Visual Analog Scale) of TEOSYAL® RHA Ultra Deep Versus Perlane-L®
Description: VAS is a 100 mm Visual Analog Scale with 0 meaning no pain and 100 meaning intolerable pain
Time Frame: During Injection and 5, 15, 30 minutes post-injection
Population: VAS are presented for the SAFT population (N=120) (see pre-assignment details) Number of patients for pain assessment after touch-up treatment are based on number of patients receiving Touch-up treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEOSYAL® RHA Ultra Deep | Perlane-L®
Number analyzed (Participants) | 120 | 120
units on a scale
  Initial injection mean pain during injection | 23.43 (21.15) | 23.85 (21.35)
  Initial injection mean pain 5 min post-injection | 6.22 (12.37) | 5.33 (12.76)
  Initial injection mean pain 15 min post-injection | 2.67 (7.38) | 2.82 (8.35)
  Initial injection mean pain 30 min post-injection | 1.83 (7.31) | 1.65 (7.61)
  Touch-up injection mean pain during injection: number analyzed (Participants) | 32 | 47
  Touch-up injection mean pain during injection | 23.63 (23.06) | 23.34 (19.32)
  Touch-up injection mean pain 5 min post-injection: number analyzed (Participants) | 32 | 47
  Touch-up injection mean pain 5 min post-injection | 8.88 (14.46) | 5.30 (8.39)
  Touch-up injection mean pain 15 min post-injection: number analyzed (Participants) | 32 | 47
  Touch-up injection mean pain 15 min post-injection | 3.56 (6.48) | 2.62 (4.88)
  Touch-up injection mean pain 30 min post-injection: number analyzed (Participants) | 32 | 47
  Touch-up injection mean pain 30 min post-injection | 1.81 (4.49) | 1.38 (3.17)

4. Secondary Outcome: Delta of the WSRS Score Between W24,36,52 and 64 and Baseline for TEOSYAL® RHA Ultra Deep Versus Perlane-L® for the Correction of Moderate to Severe NLFs Based on the Wrinkle Severity Rating Scale (WSRS) Score Assessed by the Blinded Live Evaluator (BLE)
Description: WSRS (Wrinkle Severity Rating Scale) is a validated 5-point scale with 1 being 'absent' and 5 being 'extreme'.
Time Frame: Baseline and Weeks 24, 36, 52, 64
Population: Numbers of patients analyzed correspond to patients that have completed the visits and for which data were available (See participant flow)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEOSYAL® RHA Ultra Deep | Perlane-L®
Number analyzed (Participants) | 88 | 88
units on a scale
  W24 Delta from baseline | -1.34 (0.57) | -1.16 (0.62)
  W36 Delta from baseline: number analyzed (Participants) | 86 | 86
  W36 Delta from baseline | -1.28 (0.63) | -1.12 (0.60)
  W52 Delta from baseline: number analyzed (Participants) | 77 | 77
  W52 Delta from baseline | -1.23 (0.74) | -1.05 (0.67)
  W64 Delta from baseline: number analyzed (Participants) | 65 | 65
  W64 Delta from baseline | -1.26 (0.71) | -1.11 (0.71)

5. Secondary Outcome: Delta of the WSRS Score Between W2,4,12,24,36,52,64 and Baseline for TEOSYAL® RHA Ultra Deep Versus Perlane-L® for the Correction of Moderate to Severe NLFs Based on the Wrinkle Severity Rating Scale (WSRS) Score Assessed by the Treating Investigator (TI)
Description: WSRS (Wrinkle Severity Rating Scale) is a validated 5-point scale with 1 being 'absent' and 5 being 'extreme'.
Time Frame: Baseline and Weeks 2, 4, 12, 24, 36, 52, 64
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEOSYAL® RHA Ultra Deep | Perlane-L®
Number analyzed (Participants) | 88 | 88
units on a scale
  W2 Delta from baseline | -1.77 (0.60) | -1.51 (0.68)
  W4 Delta from baseline | -1.85 (0.58) | -1.60 (0.63)
  W12 Delta from baseline | -1.70 (0.78) | -1.34 (0.74)
  W24 Delta from baseline | -1.45 (0.76) | -1.05 (0.76)
  W36 Delta from baseline: number analyzed (Participants) | 86 | 86
  W36 Delta from baseline | -1.50 (0.78) | -1.16 (0.73)
  W52 Delta from baseline: number analyzed (Participants) | 84 | 84
  W52 Delta from baseline | -1.38 (0.71) | -0.99 (0.67)
  W64 Delta from baseline | -1.32 (0.82) | -1.03 (0.77)

6. Secondary Outcome: Percentage of Responders Based on the Intra-individual Improvement of at Least One Grade in the Wrinkle Severity Rating Scale (WSRS) Compared to Baseline Assessed by the BLE
Description: A responder correspond to a subject with an intra-individual improvement of at least one grade in the WSRS compared to Baseline
Time Frame: Baseline and Weeks 24, 36, 52, 64
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | TEOSYAL® RHA Ultra Deep | Perlane-L®
Number analyzed (Participants) | 88 | 88
percentage of responders
  W24 | 97.7 [92.0 to 99.7] | 88.6 [80.1 to 94.4]
  W36: number analyzed (Participants) | 86 | 86
  W36 | 90.7 [82.5 to 95.9] | 87.2 [78.3 to 93.4]
  W52: number analyzed (Participants) | 77 | 77
  W52 | 87.0 [77.4 to 94.0] | 83.1 [72.9 to 90.7]
  W64: number analyzed (Participants) | 65 | 65
  W64 | 89.2 [79.1 to 95.6] | 84.6 [73.5 to 92.4]

7. Secondary Outcome: Percentage of Responders Based on the Intra-individual Improvement of at Least One Grade in the Wrinkle Severity Rating Scale (WSRS) Compared to Baseline Assessed by the TI
Description: as for outcome 6
Time Frame: Baseline and Weeks 2, 4, 12, 24, 36, 52, 64
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | TEOSYAL® RHA Ultra Deep | Perlane-L®
Number analyzed (Participants) | 88 | 88
percentage of responders
  W2 | 97.7 [92.0 to 99.7] | 93.2 [85.8 to 97.5]
  W4 | 100.0 [95.9 to 100.0] | 97.7 [92.0 to 99.7]
  W12 | 95.5 [88.8 to 98.8] | 88.6 [80.1 to 94.4]
  W24 | 90.9 [82.9 to 96.0] | 78.4 [68.4 to 86.5]
  W36: number analyzed (Participants) | 86 | 86
  W36 | 90.7 [82.5 to 95.9] | 83.7 [74.2 to 90.8]
  W52: number analyzed (Participants) | 84 | 84
  W52 | 92.9 [85.1 to 97.3] | 77.4 [67.0 to 85.8]
  W64: number analyzed (Participants) | 71 | 71
  W64 | 83.1 [72.3 to 91.0] | 76.1 [64.5 to 85.4]

8. Secondary Outcome: Number of Subjects Scored Either "Much Improved" or "Improved" on Global Aesthetic Improvement (GAI) by the Blinded Live Evaluator (BLE)
Description: Global Aesthetic Improvement (GAI) is a subjective 5-grade scale comprised of "much improved, improved, no change, worse, and much worse".
  GAI was assessed using the baseline photograph. Each side of the face was assessed independently.
Time Frame: Weeks 24, 36, 52, 64
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | TEOSYAL® RHA Ultra Deep | Perlane-L®
Number analyzed (Participants) | 88 | 88
Participants
  W24 | 84 | 80
  W36: number analyzed (Participants) | 86 | 86
  W36 | 80 | 77
  W52: number analyzed (Participants) | 77 | 77
  W52 | 65 | 62
  W64: number analyzed (Participants) | 65 | 65
  W64 | 52 | 47

9. Secondary Outcome: Number of Global Aesthetic Improvement (GAI) Responders (i.e., Scoring Either "Much Improved" or "Improved") on GAI Scale.
Description: Global Aesthetic Improvement (GAI) is a subjective 5-grade scale comprised of "much improved, improved, no change, worse, and much worse".
  GAI was assessed using the baseline photograph. Subjects will be instructed: "Use a mirror to compare your face to the photograph provided to you and rate the degree of aesthetic improvement by using the following scale".
  Each side of the face was assessed independently.
Time Frame: Weeks 4, 12, 24, 36, 52, 64
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | TEOSYAL® RHA Ultra Deep | Perlane-L®
Number analyzed (Participants) | 88 | 88
Participants
  W4 | 87 | 88
  W12 | 87 | 85
  W24 | 82 | 78
  W36: number analyzed (Participants) | 86 | 86
  W36 | 81 | 78
  W52: number analyzed (Participants) | 84 | 84
  W52 | 77 | 73
  W64: number analyzed (Participants) | 70 | 70
  W64 | 64 | 58

10. Secondary Outcome: Subject's Perception of Treatment Effectiveness as Per the FACE-Q (NLF Domain) Questionnaire
Description: The FACE-Q measures the experience and outcomes of aesthetic facial procedures from the patient's perspective.
  FACE-Q questionnaire is composed of 5 questions with a score linked to answers (1 being 'Not at all' and 4 being 'Extremely').
  The subject was instructed as follows: "These questions ask about how you look right now. With your nasolabial folds in mind (the deep lines that run downward from the sides of your nose), in the past week, how much have you been bothered by:", and provided response.
  * How deep your nasolabial fold are?
  * How your nasolabial folds look when your face is relaxed (still)?
  * How old your nasolabial folds make you look?
  * How your nasolabial folds look when you smile?
  * How your nasolabial folds look compared with other people your age? To calculate the FACE-Q, outcomes from all 5 questions were pooled and adapted to a scale to 100 units. Data were also transformed so that higher scores reflected a beneficial outcome.
Time Frame: Immediately post-injection, and weeks 2, 4, 12, 24, 36, 52, 64
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEOSYAL® RHA Ultra Deep | Perlane-L®
Number analyzed (Participants) | 88 | 88
units on a scale
  pre-treatment | 24.7 (19.2) | 25.7 (19.6)
  W2: number analyzed (Participants) | 87 | 87
  W2 | 77.1 (23.3) | 74.0 (23.9)
  W4 | 84.3 (21.0) | 81.2 (21.0)
  W12 | 80.1 (22.3) | 74.4 (25.0)
  W24 | 70.9 (22.3) | 66.1 (24.2)
  W36: number analyzed (Participants) | 86 | 86
  W36 | 68.9 (25.0) | 61.5 (25.5)
  W52: number analyzed (Participants) | 84 | 84
  W52 | 72.0 (25.6) | 65.9 (27.2)
  W64: number analyzed (Participants) | 70 | 70
  W64 | 69.7 (24.0) | 64.2 (27.5)

11. Secondary Outcome: Subject's Satisfaction Score
Description: Subjective 5-point scale with 1 being 'very satisfied' and 5 being 'very dissatisfied'
Time Frame: Weeks 2, 4, 12, 24, 36, 52, 64
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEOSYAL® RHA Ultra Deep | Perlane-L®
Number analyzed (Participants) | 88 | 88
units on a scale
  W2: number analyzed (Participants) | 87 | 87
  W2 | 1.49 (0.61) | 1.63 (0.88)
  W4: number analyzed (Participants) | 88 | 84
  W4 | 1.28 (0.57) | 1.31 (0.58)
  W12: number analyzed (Participants) | 87 | 84
  W12 | 1.41 (0.62) | 1.62 (0.83)
  W24: number analyzed (Participants) | 87 | 87
  W24 | 1.53 (0.66) | 1.79 (0.84)
  W36: number analyzed (Participants) | 86 | 86
  W36 | 1.64 (0.75) | 1.95 (0.96)
  W52: number analyzed (Participants) | 84 | 84
  W52 | 1.54 (0.70) | 1.77 (0.87)
  W64: number analyzed (Participants) | 70 | 70
  W64 | 1.40 (0.60) | 1.67 (0.90)

12. Secondary Outcome: Volume to Obtain Optimal Cosmetic Result (Initial Treatment + Touch-up)
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | TEOSYAL® RHA Ultra Deep | Perlane-L®
Number analyzed (Participants) | 88 | 88
mL | 1.79 (0.87) | 1.75 (0.90)

13. Secondary Outcome: Number of Subjects Receiving Touch-up Treatment
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Arm/Group | TEOSYAL® RHA Ultra Deep | Perlane-L®
Number analyzed (Participants) | 88 | 88
Participants | 28 | 38

14. Secondary Outcome: Number of Subjects Receiving Re-treatment
Time Frame: Weeks 24, 36, 52, 64
Population: Numbers of patients analyzed correspond to patients that have completed the visits (See participant flow)
Measure: Count of Participants; unit: Participants
Arm/Group | TEOSYAL® RHA Ultra Deep | Perlane-L®
Number analyzed (Participants) | 88 | 88
Participants
  W24 | 6 | 6
  W36: number analyzed (Participants) | 86 | 86
  W36 | 3 | 6
  W52: number analyzed (Participants) | 84 | 84
  W52 | 12 | 13
  W64: number analyzed (Participants) | 71 | 71
  W64 | 49 | 50

ADVERSE EVENTS:
Time Frame: 64 weeks or 68 weeks for patients receiving a re-treatment at W64
Description: The TI assessed all AEs and recorded details of seriousness, severity, duration, and action taken with study device, and relationship to the study device.
  Adverse Events are presented for the SAFT population (N=120) (see pre-assignment details)
Arm/Group | TEOSYAL® RHA Ultra Deep | Perlane-L®
Serious Adverse Events (participants affected / at risk) | 3/120 | 3/120
Other Adverse Events (participants affected / at risk) | 75/120 | 74/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TEOSYAL® RHA Ultra Deep (N=120) | Perlane-L® (N=120)
Arthralgia (General disorders) | 1 | 1 — unrelated to the study device
Diverticulitis (General disorders) | 1 | 1 — unrelated to the study device
Lung Infection (Infections and infestations) | 1 | 1 — unrelated to the study device
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TEOSYAL® RHA Ultra Deep (N=120) | Perlane-L® (N=120)
Injection Lumps/Bumps (General disorders) | 45 (52) | 34 (43)
Injection site firmness (General disorders) | 45 (52) | 34 (39)
Injection site swelling (General disorders) | 24 (28) | 17 (21)
Tenderness (General disorders) | 19 (22) | 12 (14)
Injection site discolouration (General disorders) | 13 (13) | 7 (7)
Injection site erythema (General disorders) | 8 (8) | 8 (8)
Injection site haematoma (General disorders) | 8 (8) | 4 (5)
Injection site pain (General disorders) | 6 (7) | 5 (5)
Headache (Nervous system disorders) | 6 (9) | 6 (10)
Acne (Skin and subcutaneous tissue disorders) | 5 (5) | 6 (6)
Telangiectasia (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days